CLINICAL TRIAL: NCT02499900
Title: CONFIDENCE: A Multinational, Multicenter, Randomized, Parallel Group, Open-Label Study to Assess Medication Satisfaction in Patients With Relapsing Remitting Multiple Sclerosis (RRMS) Treated With Subcutaneous Injections of Copaxone(R) (Glatiramer Acetate) 40 mg/mL Three Times a Week Compared to 20 mg/mL Daily
Brief Title: Study to Assess Medication Satisfaction in Patients With Relapsing Remitting Multiple Sclerosis Treated With Copaxone®
Acronym: CONFIDENCE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TV44400-CNS-40083; 2015-000922-12 (EudraCT Number)
Record Dates: First submitted 2015-07-01; First posted 2015-07-16 (Estimated); Results first posted 2018-08-20 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-12

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Glatiramer Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Copaxone® 40 mg/mL (Experimental): Subcutaneous Injections 40 mg/mL Three Times a Week for the core period which last 6 months. In the extension period patient are administered Copaxone® 40 mg/mL for months 7 - 12.
  Interventions: Drug: Copaxone®
- Copaxone® 20 mg/mL (Active Comparator): Subcutaneous Injections 20 mg/mL Daily for the core period which last 6 months. In the extension period patient are administered Copaxone® 40 mg/mL for months 7 - 12.
  Interventions: Drug: Copaxone®

INTERVENTIONS:
Drug: Copaxone® — Subcutaneous Injections
  Other Names: Glatiramer Acetate

SUMMARY:
The primary objective of this study is to compare patient medication satisfaction as measured by the Medication Satisfaction Questionnaire (MSQ) scores between the Copaxone 40 mg/mL three time a week (TIW) group and the Copaxone 20 mg/mL once daily (QD) group over 6 months of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women at least 18 years of age or older.
2. Patients must have a confirmed and documented RRMS diagnosis
3. Patients must be ambulatory with a Kurtzke EDSS score of 0 to 5.5 at screening visit.
4. Patients must be in a stable neurological condition, relapse-free and free of any corticosteroid treatment 30 days prior to randomization.
5. Women of child-bearing potential must have a negative urine pregnancy test at screening visit and must practice an acceptable method of birth
6. Patients must be able to sign and date a written informed consent prior to entering the study.
7. Patients must be willing and able to comply with the protocol requirements for the duration of the study.

Exclusion Criteria

1. Patient had any contraindication to Copaxone therapy.
2. Previous use of Copaxone 40 mg/mL three times per week.
3. Patients with progressive forms of MS.
4. Patients with neuromyelitis optica.
5. Use of experimental or investigational drugs, and/or participation in drug clinical studies within the 6 months prior to screening.
6. Patients who have been treated with; immunosuppressive medications, immunoglobulins and/or monoclonal antibodies, alemtuzumab, cladribine, cyclophosphamide or mitoxantrone at any time
7. Chronic (more than 30 consecutive days) systemic (IV, PO or IM) corticosteroid treatment within 6 months prior to screening visit.
8. Pregnancy or breastfeeding.
9. Clinically significant or unstable medical or surgical condition that would preclude safe and complete study participation
10. Employees of the clinical study site or any other individuals involved with the conduct of the study, or immediate family members of such individuals

    * other criteria may apply, please contact the investigator for more information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 861 (Actual)
Dates: Start 2015-08-10 (Actual); Primary Completion 2017-01-10 (Actual); Study Completion 2017-06-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (97):
- United States (15):
  - Teva Investigational Site 13485, Cullman, Alabama
  - Teva Investigational Site 13524, Carmichael, California
  - Teva Investigational Site 13478, Atlanta, Georgia
  - Teva Investigational Site 13475, Northbrook, Illinois
  - Teva Investigational Site 13472, Foxborough, Massachusetts
  - Teva Investigational Site 13479, Golden Valley, Minnesota
  - Teva Investigational Site 13483, Golden Valley, Minnesota
  - Teva Investigational Site 13487, Las Vegas, Nevada
  - Teva Investigational Site 13470, Teaneck, New Jersey
  - Teva Investigational Site 13482, New Hyde Park, New York
  - Teva Investigational Site 13471, Raleigh, North Carolina
  - Teva Investigational Site 13473, Columbus, Ohio
  - Teva Investigational Site 13477, Uniontown, Ohio
  - Teva Investigational Site 13481, Round Rock, Texas
  - Teva Investigational Site 13480, Virginia Beach, Virginia
- Argentina (3):
  - Teva Investigational Site 20061, Buenos Aires
  - Teva Investigational Site 20062, Buenos Aires
  - Teva Investigational Site 20063, Rosario
- Teva Investigational Site 33040, Vienna, Austria
- Belgium (2):
  - Teva Investigational Site 37066, Brussels
  - Teva Investigational Site 37063, Edegem
- Croatia (6):
  - Teva Investigational Site 60037, Rijeka
  - Teva Investigational Site 60039, Slavonski Brod
  - Teva Investigational Site 60034, Zagreb
  - Teva Investigational Site 60035, Zagreb
  - Teva Investigational Site 60036, Zagreb
  - Teva Investigational Site 60040, Zagreb
- Finland (2):
  - Teva Investigational Site 40014, Tampere
  - Teva Investigational Site 40015, Turku
- France (14):
  - Teva Investigational Site 35211, Besançon
  - Teva Investigational Site 35203, Bordeaux
  - Teva Investigational Site 35207, Bron
  - Teva Investigational Site 35210, Clermont-Ferrand
  - Teva Investigational Site 35208, Lille
  - Teva Investigational Site 35214, Lomme
  - Teva Investigational Site 35204, Nancy
  - Teva Investigational Site 35205, Nice
  - Teva Investigational Site 35206, Nîmes
  - Teva Investigational Site 35212, Nîmes
  - Teva Investigational Site 35213, Poissy
  - Teva Investigational Site 35202, Rennes
  - Teva Investigational Site 35201, Strasbourg
  - Teva Investigational Site 35209, Toulouse
- Germany (5):
  - Teva Investigational Site 32605, Bayreuth
  - Teva Investigational Site 32603, Dresden
  - Teva Investigational Site 32602, Hamburg
  - Teva Investigational Site 32606, Rostock
  - Teva Investigational Site 32604, Stuttgart
- Teva Investigational Site 44029, Dublin, Ireland
- Italy (8):
  - Teva Investigational Site 30169, Bari
  - Teva Investigational Site 30163, Genova
  - Teva Investigational Site 30165, Milan
  - Teva Investigational Site 30164, Milan
  - Teva Investigational Site 30161, Montichiari
  - Teva Investigational Site 30167, Naples
  - Teva Investigational Site 30166, Rome
  - Teva Investigational Site 30162, Rome
- Mexico (4):
  - Teva Investigational Site 21096, DF
  - Teva Investigational Site 21097, Mexico City
  - Teva Investigational Site 21095, Mexico City
  - Teva Investigational Site 21098, Mexico City
- Poland (12):
  - Teva Investigational Site 53352, Bydgoszcz
  - Teva Investigational Site 53354, Gdansk
  - Teva Investigational Site 53353, Gmina Końskie
  - Teva Investigational Site 53350, Katowice
  - Teva Investigational Site 53349, Kielce
  - Teva Investigational Site 53356, Lodz
  - Teva Investigational Site 53348, Lodz
  - Teva Investigational Site 53345, Lublin
  - Teva Investigational Site 53355, Olsztyn
  - Teva Investigational Site 53351, Rybnik
  - Teva Investigational Site 53347, Rzeszów
  - Teva Investigational Site 53346, Warsaw
- Teva Investigational Site 13476, Guaynabo, Puerto Rico
- Russia (12):
  - Teva Investigational Site 50392, Kaluga
  - Teva Investigational Site 50390, Kazan'
  - Teva Investigational Site 50391, Krasnoyarsk
  - Teva Investigational Site 50387, Moscow
  - Teva Investigational Site 50374, Moscow
  - Teva Investigational Site 50373, Moscow
  - Teva Investigational Site 50376, Novosibirsk
  - Teva Investigational Site 50389, Perm
  - Teva Investigational Site 50377, Saint Petersburg
  - Teva Investigational Site 50375, Saint Petersburg
  - Teva Investigational Site 50372, Tyumen
  - Teva Investigational Site 50378, Yaroslavl
- Spain (7):
  - Teva Investigational Site 31181, Burgos
  - Teva Investigational Site 31179, El Palmar
  - Teva Investigational Site 31180, Madrid
  - Teva Investigational Site 31177, Málaga
  - Teva Investigational Site 31182, Seville
  - Teva Investigational Site 31184, Seville
  - Teva Investigational Site 31178, Valencia
- Turkey (Türkiye) (4):
  - Teva Investigational Site 82052, Ankara
  - Teva Investigational Site 82051, Istanbul
  - Teva Investigational Site 82049, Istanbul
  - Teva Investigational Site 82050, Kocaeli

REFERENCES:
- [Derived] Cutter G, Veneziano A, Grinspan A, Al-Banna M, Boyko A, Zakharova M, Maida E, Pasic MB, Gandhi SK, Everts R, Cordioli C, Rossi S. Higher satisfaction and adherence with glatiramer acetate 40 mg/mL TIW vs 20 mg/mL QD in RRMS. Mult Scler Relat Disord. 2019 Aug;33:13-21. doi: 10.1016/j.msard.2019.04.036. Epub 2019 May 9. PMID 31132664

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 876 patients with RRMS were screened for enrollment into this study. Of the 876 patients screened, 861 patients at 88 centers in Russian Federation, Poland, Italy, France, Croatia, US, Mexico, Spain, Austria, Turkey, Belgium, Argentina, Germany, Finland, & Puerto Rico met entry criteria and were considered to be eligible for enrollment.
Pre-assignment Details: Of the 15 patients who were not enrolled, 2 patients were excluded on the basis of inclusion criteria not met, 4 patients were excluded on the basis of exclusion criteria met, 7 patients withdrew consent, and 2 patients were lost to follow-up before the baseline visit.
Groups:
- Copaxone® 20 mg/mL QD: Subcutaneous Injections 20 mg/mL daily (QD) for the core period which last 6 months. In the extension period patient are administered Copaxone® 40 mg/mL for months 7 - 12.
- Copaxone® 40 mg/mL TIW: Subcutaneous Injections 40 mg/mL three times a week (TIW) for the core period which last 6 months. In the extension period patient are administered Copaxone® 40 mg/mL for months 7 - 12.
Period: Core Study Period
Arm/Group | Copaxone® 20 mg/mL QD | Copaxone® 40 mg/mL TIW
Started (Intent to treat) | 430 | 431
Safety Analysis Set | 427 | 430
Completed (Completed core phase of the study) | 395 | 399
Not Completed | 35 | 32
Not completed — Other | 1 | 4
Not completed — Lost to Follow-up | 1 | 2
Not completed — Per sponsor request | 0 | 1
Not completed — Pregnancy | 1 | 0
Not completed — Protocol Violation | 3 | 0
Not completed — Withdrawal by Subject | 11 | 10
Not completed — Adverse Event | 18 | 14
Not completed — Death | 0 | 1
Period: Completed Core, Continued Into Extension
Arm/Group | Copaxone® 20 mg/mL QD | Copaxone® 40 mg/mL TIW
Started | 395 | 399
Completed | 392 | 397
Not Completed | 3 | 2
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Did not wish to take injectables drugs | 1 | 0
Not completed — Personal motivation | 1 | 0
Period: Extension Study Period
Arm/Group | Copaxone® 20 mg/mL QD | Copaxone® 40 mg/mL TIW
Started | 392 | 397
Safety Analysis Set | 392 | 396 (One participant was not treated in the Extension Study Period)
Completed | 380 | 377
Not Completed | 12 | 20
Not completed — Adverse Event | 2 | 4
Not completed — Withdrawal by Subject | 5 | 2
Not completed — Physician Decision | 2 | 5
Not completed — Pregnancy | 1 | 2
Not completed — Lost to Follow-up | 2 | 5
Not completed — Other | 0 | 2

BASELINE CHARACTERISTICS:
Population: ITT Analysis Set
Groups:
- Total: Total of all reporting groups
Arm/Group | Copaxone® 20 mg/mL QD | Copaxone® 40 mg/mL TIW | Total
Number analyzed (Participants) | 430 | 431 | 861
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.1 (10.67) | 41.0 (11.15) | 40.5 (10.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 307 | 288 | 595
  Male | 123 | 143 | 266
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 363 | 359 | 722
  Black or African American | 4 | 3 | 7
  Asian | 0 | 0 | 0
  American Indian or Alaskan Native | 1 | 0 | 1
  Native Hawaiian or Pacific Islander | 0 | 0 | 0
  Other | 59 | 63 | 122
  Missing | 3 | 6 | 9
Weight [Mean (Standard Deviation); unit: kg] — Population: Some participants were missing a baseline weight
  kg
    number analyzed (Participants) | 425 | 424 | 849
    (all) | 70.49 (16.471) | 71.85 (16.265) | 71.17 (16.373)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] — Population: Due to the missing baseline weight assessments, BMI could not be calculated for those participants.
  kg/m^2
    number analyzed (Participants) | 425 | 424 | 849
    (all) | 24.62 (5.272) | 24.93 (4.879) | 24.78 (5.079)
Height [Mean (Standard Deviation); unit: cm] — Population: Some participants were missing baseline height data.
  cm
    number analyzed (Participants) | 425 | 425 | 850
    (all) | 168.6 (9.24) | 169.4 (8.56) | 169.0 (8.91)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Medication Satisfaction Questionnaire (MSQ) to Month 6 Using a Repeated Measures ANCOVA
Description: Patient satisfaction with the study medication was assessed using the MSQ a 1-item global patient-rated scale. Patients were asked to respond on a 7-point scale, ranging from extremely dissatisfied (1) to extremely satisfied (7), to the following: "Overall, how satisfied are you with your current medication?". Positive change from baseline score indicates greater satisfaction with the medication. Estimates and p-value are obtained from baseline-adjusted repeated measures ANCOVA model with visit as a repeated effect: MSQ=baseline MSQ score+treatment+visit+treatment by visit interaction.
Time Frame: Baseline (Month 0), Months 1, 3 and 6
Population: Full analysis set (FAS) included those patients in the intent to treat (ITT) analysis set who received at least 1 dose of study drug and had at least 1 post-baseline efficacy assessment. Treatment naïve patients do not have a MSQ score at baseline so are not included.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Copaxone® 20 mg/mL QD | Copaxone® 40 mg/mL TIW
Number analyzed (Participants) | 221 | 235
units on a scale | 5.396 (0.0889) | 5.717 (0.0879)
Statistical Analysis 1: Comparison: Copaxone® 20 mg/mL QD vs Copaxone® 40 mg/mL TIW; Estimates and p-value are obtained from baseline-adjusted repeated measures ANCOVA model with visit as a repeated effect: MSQ=baseline MSQ score+treatment+visit+treatment by visit interaction. Treatment-naïve patients are not included in this analysis as MSQ is not measured at baseline for these patients; Test type: Superiority; p < 0.001, Repeated Measures ANCOVA — 0.05 level of significance; Mean Difference (Final Values) = 0.321, 95% CI 2-sided [0.1615 to 0.4814]

2. Secondary Outcome: Change From Baseline in the Treatment Satisfaction Questionnaire for Medication 9-item Version (TSQM-9) Convenience Score to Month 6 Using a Repeated Measures ANCOVA
Description: Convenience perception was measured by the 3 convenience items (items 4 to 6) within the validated TSQM-9. The responses to each of the 3 convenience items are reported on a 1-to-7 scale. The TSQM-9 convenience scale is computed, for each subject, by adding the 3 items loading on each response with the lowest possible total score (1*3 on the 3 items) subtracted from this composite score, and divided by the greatest possible score (3*7) minus the lowest possible score (3), i.e., 21-3=18. This provides a transformed score between 0 and 1 that was multiplied by 100. The final scale is 0 (Extremely Difficult/Inconvenient) to 100 (Extremely Easy/Convenient). If more than one item is missing, then the convenience scale was considered invalid for that patient. Estimates and p-value are obtained from baseline-adjusted repeated measures ANCOVA with treatment, visit, and Country/Geographical Region as main factors, visit by treatment as the interaction term, and baseline score as the covariate.
Time Frame: Baseline (Month 0), Months 1, 3 and 6
Population: Full analysis set (FAS) included those patients in the intent to treat (ITT) analysis set who received at least 1 dose of study drug and had at least 1 post-baseline efficacy assessment. Treatment naïve patients do not have TSQM-9 convenience scores at baseline and therefore are not included.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Copaxone® 20 mg/mL QD | Copaxone® 40 mg/mL TIW
Number analyzed (Participants) | 216 | 223
units on a scale | 69.740 (1.1999) | 79.189 (1.2347)
Statistical Analysis 1: Comparison: Copaxone® 20 mg/mL QD vs Copaxone® 40 mg/mL TIW; Estimates and p-value are obtained from baseline-adjusted repeated measures ANCOVA model with visit as a repeated effect: TSQM-9 convenience score=baseline TSQM-9 convenience score+treatment+CGR+treatment by visit interaction. Treatment-naïve patients are not included in this analysis as TSQM-9 is not measured at baseline for these patients; Test type: Superiority; p < 0.001, Repeated Measures ANCOVA — 0.05 level of significance; Mean Difference (Final Values) = 9.448, 95% CI 2-sided [6.9538 to 11.9429]

3. Secondary Outcome: Change From Baseline in the Modified Fatigue Impact Scale (MFIS) Total Score and Subscales to Month 6 Using a Repeated Measures ANCOVA
Description: MFIS is a modified form of the Fatigue Impact Scale based on items derived from interviews with MS patients concerning how fatigue impacts their lives. It is a structured, self-report questionnaire consisting of 21 items assessing the effects of fatigue. All 21 items are scaled 0 to 4, with higher scores indicating a greater impact of fatigue on patient's activities. The Total MFIS score ranges from 0 to 84, the Physical Subscale from 0 to 36, the Cognitive Subscale from 0 to 40, and the Psychosocial Subscale from 0 to 8. A score of 0 indicates fatigue has no impact on activities and the high-end score indicates fatigue has extreme impact on activities. Negative change from baseline values indicate improvement in the effects of fatigue. Estimates and p-values are obtained from baseline-adjusted repeated measures ANCOVA model with visit as a repeated effect: change from
Time Frame: Baseline (Month 0), Months 1, 3 and 6
Population: Full analysis set (FAS). The participant was considered invalid if any of the items were missing.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Copaxone® 20 mg/mL QD | Copaxone® 40 mg/mL TIW
Number analyzed (Participants) | 427 | 428
units on a scale
  MFIS Total Score: number analyzed (Participants) | 422 | 425
  MFIS Total Score | -2.811 (0.5166) | -3.613 (0.5052)
  MFIS Physical Subscale: number analyzed (Participants) | 422 | 425
  MFIS Physical Subscale | -1.483 (0.2599) | -1.714 (0.2535)
  MFIS Cognitive Subscale: number analyzed (Participants) | 422 | 425
  MFIS Cognitive Subscale | -0.965 (0.2553) | -1.604 (0.2503)
  MFIS Psychosocial Subscale: number analyzed (Participants) | 422 | 425
  MFIS Psychosocial Subscale | -0.306 (0.0704) | -0.204 (0.0685)
Statistical Analysis 1: Comparison: Copaxone® 20 mg/mL QD vs Copaxone® 40 mg/mL TIW; MFIS Total Score Estimates and p-values are obtained from baseline-adjusted repeated measures ANCOVA model with visit as a repeated effect: change from baseline MFIS score=baseline MFIS score+treatment+visit +CGR+treatment by visit interaction; Test type: Superiority; p = 0.208, Repeated Measures ANCOVA — 0.05 level of significance; Mean Difference (Final Values) = -0.802, 95% CI 2-sided [-2.0500 to 0.4461]
Statistical Analysis 2: Comparison: Copaxone® 20 mg/mL QD vs Copaxone® 40 mg/mL TIW; MFIS Physical Subscale Estimates and p-values are obtained from baseline-adjusted repeated measures ANCOVA model with visit as a repeated effect: change from baseline MFIS score=baseline MFIS score+treatment+visit +CGR+treatment by visit interaction; Test type: Superiority; p = 0.470, Repeated Measures ANCOVA — 0.05 level of significance; Mean Difference (Final Values) = -0.231, 95% CI 2-sided [-0.8588 to 0.3962]
Statistical Analysis 3: Comparison: Copaxone® 20 mg/mL QD vs Copaxone® 40 mg/mL TIW; MFIS Cognitive Subscale Estimates and p-values are obtained from baseline-adjusted repeated measures ANCOVA model with visit as a repeated effect: change from baseline MFIS score=baseline MFIS score+treatment+visit +CGR+treatment by visit interaction; Test type: Superiority; p = 0.043, Repeated Measures ANCOVA — 0.05 level of significance; Mean Difference (Final Values) = -0.639, 95% CI 2-sided [-1.2564 to -0.0214]
Statistical Analysis 4: Comparison: Copaxone® 20 mg/mL QD vs Copaxone® 40 mg/mL TIW; MFIS Psychosocial Subscale Estimates and p-values are obtained from baseline-adjusted repeated measures ANCOVA model with visit as a repeated effect: change from baseline MFIS score=baseline MFIS score+treatment+visit +CGR+treatment by visit interaction; Test type: Superiority; p = 0.237, Repeated Measures ANCOVA — 0.05 level of significance; Mean Difference (Final Values) = 0.102, 95% CI 2-sided [-0.0672 to 0.2711]

4. Secondary Outcome: Change From Baseline in the Mental Health Index (MHI) Total Score and Subscales to Month 6 Using a Repeated Measures ANCOVA
Description: The MHI consists of 18 items and provides an assessment of 4 subscales of mental health, including Anxiety (5 items), Depression (4 items), Behavioral control (4 items), and Positive Affect (4 items), and 1 Total Score. The subscales and Total Score for analyses range from 0 to 100, with 0 indicating not mentally healthy and 100 indicating superior mental health. Positive change from baseline scores indicate improved mental health. Estimates and p-values are obtained from baseline-adjusted repeated measures ANCOVA model with visit as a repeated effect: change from baseline MHI score=baseline MHI Total Score +treatment +visit +country/geographic region +treatment by visit interaction. If a participant skipped x items of y items, the scale was not computed: - MHI Total Score - 9 of 19 - Anxiety subscale - 2 of 5 - Depression subscale - 2 of 4 - Behavioral Control subscale - 2 of 4 - MHI Positive Affect subscale - 2 of 4
Time Frame: Baseline (Month 0), Months 1, 3 and 6
Population: Full analysis set.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Copaxone® 20 mg/mL QD | Copaxone® 40 mg/mL TIW
Number analyzed (Participants) | 427 | 428
units on a scale
  MHI Total Score | 3.136 (0.5381) | 3.842 (0.5249)
  Anxiety subscale | 5.468 (0.6861) | 5.609 (0.6695)
  Depression subscale | 3.773 (0.6433) | 4.253 (0.6270)
  Behavioral Control subscale: number analyzed (Participants) | 423 | 428
  Behavioral Control subscale | 0.659 (0.6133) | 2.526 (0.6000)
  MHI Positive Affect subscale: number analyzed (Participants) | 423 | 428
  MHI Positive Affect subscale | 3.024 (0.7306) | 2.932 (0.7126)
Statistical Analysis 1: Comparison: Copaxone® 20 mg/mL QD vs Copaxone® 40 mg/mL TIW; Total Score Estimates and p-values are obtained from baseline-adjusted repeated measures ANCOVA model with visit as a repeated effect: change from baseline MHI score=baseline MHI Total Score +treatment +visit +country/geographic region +treatment by visit interaction; Test type: Superiority; p = 0.287, Repeated Measures ANCOVA — 0.05 level of significance; Mean Difference (Final Values) = 0.706, 95% CI 2-sided [-0.5947 to 1.0074]
Statistical Analysis 2: Comparison: Copaxone® 20 mg/mL QD vs Copaxone® 40 mg/mL TIW; Anxiety subscale Estimates and p-values are obtained from baseline-adjusted repeated measures ANCOVA model with visit as a repeated effect: change from baseline MHI score=baseline MHI Total Score +treatment +visit +country/geographic region +treatment by visit interaction; Test type: Superiority; p = 0.868, Repeated Measures ANCOVA — 0.05 level of significance; Mean Difference (Final Values) = 0.141, 95% CI 2-sided [-1.5179 to 1.7991]
Statistical Analysis 3: Comparison: Copaxone® 20 mg/mL QD vs Copaxone® 40 mg/mL TIW; Depression subscale estimates and p-values are obtained from baseline-adjusted repeated measures ANCOVA model with visit as a repeated effect: change from baseline MHI score=baseline MHI Total Score +treatment +visit +country/geographic region +treatment by visit interaction; Test type: Superiority; p = 0.544, Repeated Measures ANCOVA — 0.05 level of significance; Mean Difference (Final Values) = 0.481, 95% CI 2-sided [-1.0734 to 2.0348]
Statistical Analysis 4: Comparison: Copaxone® 20 mg/mL QD vs Copaxone® 40 mg/mL TIW; Behavioral Control subscale Estimates and p-values are obtained from baseline-adjusted repeated measures ANCOVA model with visit as a repeated effect: change from baseline MHI score=baseline MHI Total Score +treatment +visit +country/geographic region +treatment by visit interaction; Test type: Superiority; p = 0.014, Repeated Measures ANCOVA — 0.05 level of significance; Mean Difference (Final Values) = 1.867, 95% CI 2-sided [0.3843 to 3.3487]
Statistical Analysis 5: Comparison: Copaxone® 20 mg/mL QD vs Copaxone® 40 mg/mL TIW; MHI Positive Affect subscale Estimates and p-values are obtained from baseline-adjusted repeated measures ANCOVA model with visit as a repeated effect: change from baseline MHI score=baseline MHI Total Score +treatment +visit +country/geographic region +treatment by visit interaction; Test type: Superiority; p = 0.919, Repeated Measures ANCOVA — 0.05 level of significance; Mean Difference (Final Values) = -0.092, 95% CI 2-sided [-1.8565 to 1.6728]

5. Secondary Outcome: Change From Baseline in the Beck Depression Inventory II (BDI-II) Total Score to Month 6 Using a Repeated Measures ANCOVA
Description: Depressive symptoms were measured by the BDI-II, a 21-item, self-reported rating inventory that measures characteristic attitudes and symptoms of depression. The BDI-II assesses mood, pessimism, sense of failure, self-dissatisfaction, guilt, punishment, self-dislike, self-accusation, suicidal ideas, sadness, crying, irritability, social withdrawal, body image, work difficulties, insomnia, fatigue, appetite, weight loss, bodily preoccupation, and loss of libido. Each of the 21 items is rated on a 4-point scale ranging from 0 to 3. BDI-II Total Score indicates the severity of depression and has a total range of 0 to 63. For those clinically diagnosed, scores from 0-13 represent minimal depressive symptoms, scores of 14-19 indicate mild depression, scores of 20-28 indicate moderate depression, and scores of 30-63 indicate severe depression. Negative change from baseline scores indicate improvement.
Time Frame: Baseline (Month 0), Months 1, 3 and 6
Population: Full analysis set.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Copaxone® 20 mg/mL QD | Copaxone® 40 mg/mL TIW
Number analyzed (Participants) | 422 | 426
units on a scale | -1.525 (0.2560) | -1.585 (0.2495)
Statistical Analysis 1: Comparison: Copaxone® 20 mg/mL QD vs Copaxone® 40 mg/mL TIW; Estimates and p-values are obtained from baseline-adjusted repeated measures ANCOVA model with visit as a repeated effect: change from baseline BDI-II total score=baseline BDI-II total score+treatment+visit+country/geographic region +treatment by visit interaction; Test type: Superiority; p = 0.851, Repeated Measures ANCOVA — 0.05 level of significance; Mean Difference (Final Values) = -0.059, 95% CI 2-sided [-0.6777 to 0.5592]

6. Secondary Outcome: Participants With Treatment-Emergent Adverse Events (TEAEs) During Both the Core Period and Extension Periods
Description: An adverse event (AE) is defined as any study-related event that represents a change (positive or negative) in frequency or severity from a baseline (prestudy) event (if any), regardless of the presence of causal relationship or medical significance. Treatment-emergent adverse events are defined as any adverse event with a start date on or after the first study dose date. The investigator determined relation to study drug. A severe AE is defined as an inability to carry out usual activities. A serious AE (SAE) is defined by federal regulation as any AE occurring at any dose that results in any of the following outcomes: death, life-threatening AE, hospitalization or prolongation of existing hospitalization, a persistent or significant disability/incapacity, or a congenital anomaly/birth defect. Although a subject may have had 2 or more adverse experiences the subject is counted only once in a category. The same subject may appear in different categories.
Time Frame: Core: Day 1 to Month 6 Extension: Month 7 to Month 12
Population: Safety population
Measure: Count of Participants; unit: Participants
Groups:
- Copaxone® 20 mg/mL QD (Core): Subcutaneous injections of Copaxone 20 mg/mL daily (QD) for the core period from Day 1 to Month 6.
- Copaxone® 40 mg/mL TIW (Core): Subcutaneous injections of Copaxone 40 mg/mL three times a week (TIW) for the core period from Day 1 to Month 6.
- Copaxone® 40 mg/mL TIW (Switch-Extension): Participants who were administered daily Copaxone 20 mg/mL daily injections during the core period, were switched to 40 mg/mL three times a week (TIW) injections for the extension period (Months 7-12)
- Copaxone® 40 mg/mL TIW (Extension): Participants who were administered Copaxone 40 mg/mL three times a week (TIW) injections during the core period, continued Copaxone at that same dosage for the extension period (Months 7-12)
Arm/Group | Copaxone® 20 mg/mL QD (Core) | Copaxone® 40 mg/mL TIW (Core) | Copaxone® 40 mg/mL TIW (Switch-Extension) | Copaxone® 40 mg/mL TIW (Extension)
Number analyzed (Participants) | 427 | 430 | 392 | 396
Participants
  >=1 TEAE | 219 | 231 | 132 | 129
  >= 1 serious TEAE | 8 | 13 | 3 | 2
  >=1 serious fatal TEAE | 0 | 0 | 0 | 0
  >=1 serious and related TEAE | 1 | 2 | 0 | 0
  >=1 Severe TEAE | 4 | 3 | 1 | 0
  >=1 injection-related TEAE | 149 | 146 | 38 | 25
  >=1 TEAE leading to withdrawal | 18 | 13 | 2 | 3

ADVERSE EVENTS:
Time Frame: - Core study period: Day 1 to Month 6 - Extension study period: Month 7 to Month 12
Arm/Group | Copaxone® 20 mg/mL QD (Core) | Copaxone® 40 mg/mL TIW (Core) | Copaxone® 40 mg/mL TIW (Switch-Extension) | Copaxone® 40 mg/mL TIW (Extension)
All-Cause Mortality (participants affected / at risk) | 0/427 | 1/430 | 0/392 | 0/396
Serious Adverse Events (participants affected / at risk) | 8/427 | 13/430 | 3/392 | 2/396
Other Adverse Events (participants affected / at risk) | 121/427 | 117/430 | 22/392 | 15/396
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Copaxone® 20 mg/mL QD (Core) (N=427) | Copaxone® 40 mg/mL TIW (Core) (N=430) | Copaxone® 40 mg/mL TIW (Switch-Extension) (N=392) | Copaxone® 40 mg/mL TIW (Extension) (N=396)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pituitary hyperplasia (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Escherichia sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intentional overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Scapula fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Multiple sclerosis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Multiple sclerosis relapse (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Uterine polyp (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Copaxone® 20 mg/mL QD (Core) (N=427) | Copaxone® 40 mg/mL TIW (Core) (N=430) | Copaxone® 40 mg/mL TIW (Switch-Extension) (N=392) | Copaxone® 40 mg/mL TIW (Extension) (N=396)
Injection site bruising (General disorders) | 24 (24) | 17 (17) | 5 (5) | 4 (4)
Injection site erythema (General disorders) | 71 (75) | 61 (65) | 10 (10) | 4 (4)
Injection site haemorrhage (General disorders) | 20 (23) | 22 (26) | 2 (2) | 3 (3)
Injection site pain (General disorders) | 84 (92) | 89 (109) | 10 (11) | 5 (6)
Injection site pruritus (General disorders) | 58 (61) | 37 (40) | 5 (5) | 4 (4)
Injection site swelling (General disorders) | 34 (34) | 32 (32) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
This study's 'interim' CSR covered the Core Period and used a cut-off date. The 'final' CSR covered the entire study. AE counts as reported here reflect the entire database and show minor differences from the interim CSR due to the cut-off date.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.